CLINICAL TRIAL: NCT06058000
Title: A Phase 2, Randomized, Double-blind,Placebo Controlled, Parallel Group Study to Assess Efficacy, Safety, and Pharmacokinetics (PK) of QLM3003 Ointment in Participants With Mild or Moderate Atopic Dermatitis
Brief Title: A Phase 2 Study of QLM3003 Ointment in Participants With Mild or Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLM3003-201
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- QLM3003 Low Dose (Experimental): 2% cream applied once daily (QD)
  Interventions: Drug: 2% QLM3003
- QLM3003 Middle Dose (Experimental): 1.5% cream applied twice daily (BID)
  Interventions: Drug: 1.5% QLM3003
- QLM3003 High Dose (Experimental): 2% cream applied twice daily (BID)
  Interventions: Drug: 2% QLM3003
- Placebo Comparator: Vehicle (Placebo Comparator): Vehicle cream applied twice daily (BID)
  Interventions: Drug: Vehicle (Placebo)
- High Placebo Comparator: Vehicle (Placebo Comparator): Vehicle cream applied twice daily (BID)
  Interventions: Drug: Vehicle (Placebo)

INTERVENTIONS:
Drug: 1.5% QLM3003 — QLM3003 topical cream
  Arms: QLM3003 Middle Dose
Drug: 2% QLM3003 — QLM3003 topical cream
  Arms: QLM3003 High Dose; QLM3003 Low Dose
Drug: Vehicle (Placebo) — Vehicle topical cream
  Arms: High Placebo Comparator: Vehicle; Placebo Comparator: Vehicle

SUMMARY:
The purpose of this study is to assess efficacy, safety, and pharmacokinetics (PK) of QLM3003 Ointment in participants with mild or moderate atopic dermatitis.

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, double-blind,placebo controlled, parallel group study to assess efficacy, safety, and pharmacokinetics (PK) of QLM3003 Ointment in participants with mild or moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* The subjects understand and comply with the study requirements, voluntarily participate in the study and sign the informed consent form.
* Ages at ≥18 and ≤ 65 years.
* The diagnosis of atopic dermatitis will be confirmed according to the criteria of Hanifin and Rajka at the Screening Visit and Have a clinical diagnosis of atopic dermatitis for at least 6 months.
* Have an Investigator's Global Assessment (IGA) score of 2, or3 at screening and at baseline.
* Have atopic dermatitis on the head (excluding hair-bearing scalp), neck, trunk, or limbs, covering at least 2% of total BSA and up to and including 20% of total BSA at Screening and at baseline.

Exclusion Criteria:

* Subjects with other dermatologic disease besides AD whose presence or treatments could interfere the assessment of disease (eg, psoriasis).
* In the opinion of the investigator, have any clinically significant laboratory abnormality that would affect the participant's participation in the study.
* Use of topical treatments for AD within 2 weeks of baseline.
* Vaccinated or exposed to a live or attenuated vaccine within the 12 weeks of baseline, or is expected to be vaccinated these vaccines during treatment.
* A history of alcohol or substance abuse within 12 months prior to Screening that in the opinion of the investigator will preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving >=75% Improvement in Eczema Area and Severity Index Total Score (EASI-75) From Baseline at Weeks 8 | Baseline, Weeks 8
  EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each 4 body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Investigator's Global Assessment (IGA) Score Clear (0) or Almost Clear (1) and a Reduction From Baseline of Greater Than or Equal to ( >=2) Points at Week 8 | Baseline, Weeks 8
  IGA assesses severity of participant's AD on a 5 point scale. 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting and 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Higher scores indicating more severity of AD. Assessment excluded soles, palms and scalp.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Doctor, Principal Investigator — First Hospital of China Medical University; Furen zhang, Doctor, Principal Investigator — Dermatology Hospital of Shandong First Medical University
Locations (2):
- China (2):
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Dermatology Hospital of Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No